CLINICAL TRIAL: NCT06881069
Title: Reach Through Equitable Implementation in Utah (REI-UT)
Brief Title: Reach Through Equitable Implementation in Utah
Acronym: REI-UT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: HCI165288; 5U54CA280812-02 (NIH)
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Tobacco Use Cessation; Tobacco Use; Tobacco Smoking; Tobacco Chewing; Tobacco Dependence
MeSH Terms: conditions — Tobacco Use Cessation; Tobacco Use; Tobacco Smoking; Tobacco Use Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (21):
- 1: Clinic Level Intervention Only (Other): Patients who enrolled in Quit Services within 4 weeks after the clinical encounter will not be randomized to patient level conditions.
  Clinic Level: AAC - Tobacco, AAC - SDOH Bundled/Non-Bundled: NA PRN/RPN: NA Dose: NA
  Interventions: Behavioral: Clinic Level: AAC - SDOH, AAC - Tobacco
- 2: Non-Bundled, RPN, CA1 (Experimental): Patients who do not enroll Quit Services within 4 weeks after their clinical encounter will be randomized to receive patient-level strategies.
  Patients will receive a single proactive outreach from the CA (CA1) with content that focuses solely on enrolling in Quit Services (Non-Bundled), and will have the opportunity to request calls from a patient navigator (RPN).
  Bundled/Non-Bundled: Non-Bundled PRN/RPN: RPN Dose: CA1
  Interventions: Behavioral: Non-Bundled; Behavioral: Dose 1; Behavioral: RPN
- 3: Non-Bundled, RPN, CA3 (Experimental): Patients who do not enroll Quit Services within 4 weeks of their clinical encounter will be randomized to receive patient-level strategies.
  Patients will receive three proactive outreach opportunities from the CA (CA3) with content that focuses solely on enrolling in Quit Services (Non-Bundled), and will have the opportunity to request calls from a patient navigator (RPN).
  Bundled/Non-Bundled: Non-Bundled PRN/RPN: RPN Dose: CA3
  Interventions: Behavioral: Non-Bundled; Behavioral: Dose 3; Behavioral: RPN
- 4: Non-Bundled, RPN, CA6 (Experimental): Patients who do not enroll Quit Services within 4 weeks of their clinical encounter will be randomized to receive patient-level strategies.
  Patients will receive six proactive outreach opportunities from the CA (CA6) with content that focuses solely on enrolling in Quit Services (Non-Bundled), and will have the opportunity to request calls from a patient navigator (RPN).
  Bundled/Non-Bundled: Non-Bundled PRN/RPN: RPN Dose: CA6
  Interventions: Behavioral: Non-Bundled; Behavioral: Dose 6; Behavioral: RPN
- 5: Non-Bundled, RPN, CA9 (Experimental): Patients who do not enroll Quit Services within 4 weeks of their clinical encounter will be randomized to receive patient-level strategies.
  Patients will receive nine proactive outreach opportunities from the CA (CA9) with content that focuses solely on enrolling in Quit Services (Non-Bundled), and will have the opportunity to request calls from a patient navigator (RPN).
  Bundled/Non-Bundled: Non-Bundled PRN/RPN: RPN Dose: CA9
  Interventions: Behavioral: Non-Bundled; Behavioral: Dose 9; Behavioral: RPN
- 6: Non-Bundled, RPN, CA12 (Experimental): Patients who do not enroll Quit Services within 4 weeks of their clinical encounter will be randomized to receive patient-level strategies.
  Patients will receive twelve proactive outreach opportunities from the CA (CA12) with content that focuses solely on enrolling in Quit Services (Non-Bundled), and will have the opportunity to request calls from a patient navigator (RPN).
  Bundled/Non-Bundled: Non-Bundled PRN/RPN: RPN Dose: CA12
  Interventions: Behavioral: Non-Bundled; Behavioral: Dose 12; Behavioral: RPN
- 7: Non-Bundled, PPN Dose, CA1 (Experimental): Patients who do not enroll Quit Services within 4 weeks of their clinical encounter will be randomized to receive patient-level strategies.
  Patients will receive one proactive outreach opportunity from the CA (CA1) with content that focuses solely on enrolling in Quit Services (Non-Bundled), and will receive proactive calls from a patient navigator (PPN).
  Bundled/Non-Bundled: Non-Bundled PRN/RPN: PPN Dose: CA1
  Interventions: Behavioral: Non-Bundled; Behavioral: Dose 1; Behavioral: PPN
- 8: Non-Bundled, PPN Dose, CA3 (Experimental): Patients who do not enroll Quit Services within 4 weeks of their clinical encounter will be randomized to receive patient-level strategies.
  Patients will receive three proactive outreach opportunities from the CA (CA3) with content that focuses solely on enrolling in Quit Services (Non-Bundled), and will receive proactive calls from a patient navigator (PPN).
  Bundled/Non-Bundled: Non-Bundled PRN/RPN: PPN Dose: CA3
  Interventions: Behavioral: Non-Bundled; Behavioral: Dose 3; Behavioral: PPN
- 9: Non-Bundled, PPN Dose, CA6 (Experimental): Patients who do not enroll Quit Services within 4 weeks of their clinical encounter will be randomized to receive patient-level strategies.
  Patients will receive six proactive outreach opportunities from the CA (CA6) with content that focuses solely on enrolling in Quit Services (Non-Bundled), and will receive proactive calls from a patient navigator (PPN).
  Bundled/Non-Bundled: Non-Bundled PRN/RPN: PPN Dose: CA6
  Interventions: Behavioral: Non-Bundled; Behavioral: Dose 6; Behavioral: PPN
- 10: Non-Bundled, PPN Dose, CA9 (Experimental): Patients who do not enroll Quit Services within 4 weeks of their clinical encounter will be randomized to receive patient-level strategies.
  Patients will receive nine proactive outreach opportunities from the CA (CA9) with content that focuses solely on enrolling in Quit Services (Non-Bundled), and will receive proactive calls from a patient navigator (PPN).
  Bundled/Non-Bundled: Non-Bundled PRN/RPN: PPN Dose: CA9
  Interventions: Behavioral: Non-Bundled; Behavioral: Dose 9; Behavioral: PPN
- 11: Non-Bundled, PPN Dose, CA12 (Experimental): Patients who do not enroll Quit Services within 4 weeks of their clinical encounter will be randomized to receive patient-level strategies.
  Patients will receive twelve proactive outreach opportunities from the CA (CA12) with content that focuses solely on enrolling in Quit Services (Non-Bundled), and will receive proactive calls from a patient navigator (PPN).
  Bundled/Non-Bundled: Non-Bundled PRN/RPN: PPN Dose: CA12
  Interventions: Behavioral: Non-Bundled; Behavioral: Dose 12; Behavioral: PPN
- 12: Bundled, RPN, CA1 (Experimental): Patients who do not enroll Quit Services within 4 weeks of their clinical encounter will be randomized to receive patient-level strategies.
  Patients will receive one proactive outreach opportunity from the CA (CA1) with content that focuses on enrolling in Quit Services and addressing SDOH (Bundled), and will have the opportunity to request calls from a patient navigator (RPN).
  Bundled/Non-Bundled: Bundled PRN/RPN: RPN Dose: CA1
  Interventions: Behavioral: Bundled; Behavioral: Dose 1; Behavioral: RPN
- 13: Bundled, RPN, CA3 (Experimental): Patients who do not enroll Quit Services within 4 weeks of their clinical encounter will be randomized to receive patient-level strategies.
  Patients will receive three proactive outreach opportunities from the CA (CA3) with content that focuses on enrolling in Quit Services and addressing SDOH (Bundled), and will have the opportunity to request calls from a patient navigator (RPN).
  Bundled/Non-Bundled: Bundled PRN/RPN: RPN Dose: CA3
  Interventions: Behavioral: Bundled; Behavioral: Dose 3; Behavioral: RPN
- 14: Bundled, RPN, CA6 (Experimental): Patients who do not enroll Quit Services within 4 weeks of their clinical encounter will be randomized to receive patient-level strategies.
  Patients will receive six proactive outreach opportunities from the CA (CA6) with content that focuses on enrolling in Quit Services and addressing SDOH (Bundled), and will have the opportunity to request calls from a patient navigator (RPN).
  Bundled/Non-Bundled: Bundled PRN/RPN: RPN Dose: CA6
  Interventions: Behavioral: Bundled; Behavioral: Dose 6; Behavioral: RPN
- 15: Bundled, RPN, CA9 (Experimental): Patients who do not enroll Quit Services within 4 weeks of their clinical encounter will be randomized to receive patient-level strategies.
  Patients will receive nine proactive outreach opportunities from the CA (CA9) with content that focuses on enrolling in Quit Services and addressing SDOH (Bundled), and will have the opportunity to request calls from a patient navigator (RPN).
  Bundled/Non-Bundled: Bundled PRN/RPN: RPN Dose: CA9
  Interventions: Behavioral: Bundled; Behavioral: Dose 9; Behavioral: RPN
- 16: Bundled, RPN, CA12 (Experimental): Patients who do not enroll Quit Services within 4 weeks of their clinical encounter will be randomized to receive patient-level strategies.
  Patients will receive 12 proactive outreach opportunities from the CA (CA12) with content that focuses on enrolling in Quit Services and addressing SDOH (Bundled), and will have the opportunity to request calls from a patient navigator (RPN).
  Bundled/Non-Bundled: Bundled PRN/RPN: RPN Dose: CA12
  Interventions: Behavioral: Bundled; Behavioral: Dose 12; Behavioral: RPN
- 17: Bundled, PPN, CA1 (Experimental): Patients who do not enroll Quit Services within 4 weeks of their clinical encounter will be randomized to receive patient-level strategies.
  Patients will receive one proactive outreach opportunity from the CA (CA1) with content that focuses on enrolling in Quit Services and addressing SDOH (Bundled), and will receive proactive calls from a patient navigator (PPN).
  Bundled/Non-Bundled: Bundled PRN/RPN: PPN Dose: CA1
  Interventions: Behavioral: Bundled; Behavioral: Dose 1; Behavioral: PPN
- 18: Bundled, PPN, CA3 (Experimental): Patients who do not enroll Quit Services within 4 weeks of their clinical encounter will be randomized to receive patient-level strategies.
  Patients will receive three proactive outreach opportunities from the CA (CA3) with content that focuses on enrolling in Quit Services and addressing SDOH (Bundled), and will receive proactive calls from a patient navigator (PPN).
  Bundled/Non-Bundled: Bundled PRN/RPN: PPN Dose: CA3
  Interventions: Behavioral: Bundled; Behavioral: Dose 3; Behavioral: PPN
- 19: Bundled, PPN, CA6 (Experimental): Patients who do not enroll Quit Services within 4 weeks of their clinical encounter will be randomized to receive patient-level strategies.
  Patients will receive six proactive outreach opportunities from the CA (CA6) with content that focuses on enrolling in Quit Services and addressing SDOH (Bundled), and will receive proactive calls from a patient navigator (PPN).
  Bundled/Non-Bundled: Bundled PRN/RPN: PPN Dose: CA6
  Interventions: Behavioral: Bundled; Behavioral: Dose 6; Behavioral: PPN
- 20: Bundled, PPN, CA9 (Experimental): Patients who do not enroll Quit Services within 4 weeks of their clinical encounter will be randomized to receive patient-level strategies.
  Patients will receive nine proactive outreach opportunities from the CA (CA9) with content that focuses on enrolling in Quit Services and addressing SDOH (Bundled), and will receive proactive calls from a patient navigator (PPN).
  Bundled/Non-Bundled: Bundled PRN/RPN: PPN Dose: CA9
  Interventions: Behavioral: Bundled; Behavioral: Dose 9; Behavioral: PPN
- 21: Bundled, PPN, CA12 (Experimental): Patients who do not enroll Quit Services within 4 weeks of their clinical encounter will be randomized to receive patient-level strategies.
  Patients will receive twelve proactive outreach opportunities from the CA (CA12) with content that focuses on enrolling in Quit Services and addressing SDOH (Bundled), and will receive proactive calls from a patient navigator (PPN).
  Bundled/Non-Bundled: Bundled PRN/RPN: PPN Dose: CA12
  Interventions: Behavioral: Bundled; Behavioral: Dose 12; Behavioral: PPN

INTERVENTIONS:
Behavioral: Clinic Level: AAC - SDOH, AAC - Tobacco — Ask-Advise-Connect (AAC) is a health information technology (HIT) implementation strategy that consists of EHR-based point-of-care supports for the assessment of tobacco use and Social Drivers of Health (SDOH).
  Arms: 1: Clinic Level Intervention Only
Behavioral: Non-Bundled — All patient level strategies will address only the content of increasing reach of the Utah Tobacco Quit Services.
  Arms: 10: Non-Bundled, PPN Dose, CA9; 11: Non-Bundled, PPN Dose, CA12; 2: Non-Bundled, RPN, CA1; 3: Non-Bundled, RPN, CA3; 4: Non-Bundled, RPN, CA6; 5: Non-Bundled, RPN, CA9; 6: Non-Bundled, RPN, CA12; 7: Non-Bundled, PPN Dose, CA1; 8: Non-Bundled, PPN Dose, CA3; 9: Non-Bundled, PPN Dose, CA6
Behavioral: Bundled — All patient level strategies will address the content of increasing reach of the Utah Tobacco Quit Services and SDOH.
  Arms: 12: Bundled, RPN, CA1; 13: Bundled, RPN, CA3; 14: Bundled, RPN, CA6; 15: Bundled, RPN, CA9; 16: Bundled, RPN, CA12; 17: Bundled, PPN, CA1; 18: Bundled, PPN, CA3; 19: Bundled, PPN, CA6; 20: Bundled, PPN, CA9; 21: Bundled, PPN, CA12
Behavioral: Dose 1 — The number of proactive outreach opportunities for CA the patient receives. Patient will receive 1 opportunity for CA, over 12 months following a patient's initial clinic visit, that includes a simple one-touch response to directly connect to the Quit Services or the CHW.
  Arms: 12: Bundled, RPN, CA1; 17: Bundled, PPN, CA1; 2: Non-Bundled, RPN, CA1; 7: Non-Bundled, PPN Dose, CA1
Behavioral: Dose 3 — The number of proactive outreach opportunities for CA the patient receives. Patient will receive 3 opportunities for CA, over 12 months following a patient's initial clinic visit, that includes a simple one-touch response to directly connect to the Quit Services or the CHW.
  Arms: 13: Bundled, RPN, CA3; 18: Bundled, PPN, CA3; 3: Non-Bundled, RPN, CA3; 8: Non-Bundled, PPN Dose, CA3
Behavioral: Dose 6 — The number of proactive outreach opportunities for CA the patient receives. Patient will receive 6 opportunities for CA, over 12 months following a patient's initial clinic visit, that includes a simple one-touch response to directly connect to the Quit Services or the CHW.
  Arms: 14: Bundled, RPN, CA6; 19: Bundled, PPN, CA6; 4: Non-Bundled, RPN, CA6; 9: Non-Bundled, PPN Dose, CA6
Behavioral: Dose 9 — The number of proactive outreach opportunities for CA the patient receives. Patient will receive 9 opportunities for CA, over 12 months following a patient's initial clinic visit, that includes a simple one-touch response to directly connect to the Quit Services or the CHW.
  Arms: 10: Non-Bundled, PPN Dose, CA9; 15: Bundled, RPN, CA9; 20: Bundled, PPN, CA9; 5: Non-Bundled, RPN, CA9
Behavioral: Dose 12 — The number of proactive outreach opportunities for CA the patient receives. Patient will receive 12 opportunities for CA, over 12 months following a patient's initial clinic visit, that includes a simple one-touch response to directly connect to the Quit Services or the CHW.
  Arms: 11: Non-Bundled, PPN Dose, CA12; 16: Bundled, RPN, CA12; 21: Bundled, PPN, CA12; 6: Non-Bundled, RPN, CA12
Behavioral: RPN — Reactive Patient Navigation Only (RPN): Patient can request to speak to a CHW, over 12 months following a patient's initial clinic visit, at any time.
  Arms: 12: Bundled, RPN, CA1; 13: Bundled, RPN, CA3; 14: Bundled, RPN, CA6; 15: Bundled, RPN, CA9; 16: Bundled, RPN, CA12; 2: Non-Bundled, RPN, CA1; 3: Non-Bundled, RPN, CA3; 4: Non-Bundled, RPN, CA6; 5: Non-Bundled, RPN, CA9; 6: Non-Bundled, RPN, CA12
Behavioral: PPN — Proactive Patient Navigation (PPN): Patient is proactively called, over 12 months following a patient's initial clinic visit, by a CHW up to 4 times.
  Arms: 10: Non-Bundled, PPN Dose, CA9; 11: Non-Bundled, PPN Dose, CA12; 17: Bundled, PPN, CA1; 18: Bundled, PPN, CA3; 19: Bundled, PPN, CA6; 20: Bundled, PPN, CA9; 21: Bundled, PPN, CA12; 7: Non-Bundled, PPN Dose, CA1; 8: Non-Bundled, PPN Dose, CA3; 9: Non-Bundled, PPN Dose, CA6

SUMMARY:
The goal of this pragmatic, multilevel Type III Hybrid Effectiveness-Implementation trial is to increase the reach of existing evidence-based interventions (EBIs) for tobacco cessation and to mitigate the impact of adverse Social Drivers of Health (SDOH) among safety-net healthcare system patients who live in persistent poverty (PP) census tracts.

Aim 1: Test the ability of patient-level Conversational Agents (CA) & Patient Navigation (PN) dissemination strategies to increase the Reach (primary outcome) of evidence-based tobacco cessation treatment delivered via the Utah Tobacco and Nicotine Quit Services (Quit Services) among Community Health Center (CHC) patients who use tobacco and live in persistent poverty census tracts. Secondary analyses will examine the outcome of Reach of services for SDOH among these patients and will evaluate both 1) patient-level CA and PN dissemination strategies and 2) a clinic-level implementation strategy using a pre-post design.

Aim 2: Explore contextual factors (e.g., clinic size, patient composition, rurality, patient demographics) related to the Reach, Adoption, Implementation, and potential Maintenance of strategies.

Aim 3: Determine the cost-effectiveness of clinic and patient-level strategies based on Quit Services enrollment and service receipt for SDOH.

This trial implements a clinic-level implementation strategy, Ask-Advise-Connect (AAC), to address tobacco cessation and needs around social drivers of health for patients in all participating clinics. Eligible patients who are not enrolled in Quit Services four weeks after the clinical encounter, will receive text messages from a chatbot offering information and connections to the Quit Services and patient navigation support from a Community Health Worker.

DETAILED DESCRIPTION:
REI-UT is a pragmatic, multilevel Type III Hybrid Effectiveness-Implementation trial with a 2x2x5 factorial experimental design. It consists of clinic level implementation strategies (AAC - SDOH, AAC - Tobacco), which will be implemented in all participating clinics and four patient level interventions, which will be randomized based on Quit Services response. Individuals who do not enroll in the Quit Services after four weeks of receiving the clinic level strategy will be randomly assigned to one of 20 conditions in the 2X2X5 factorial design.

Clinic Level Implementation Strategy:

Ask-Advise-Connect (AAC) is a health information technology (HIT) implementation strategy that consists of Electronic Health Record (EHR) based point of care supports for the assessment of and referral to resources for tobacco use and SDOH (ASK).

Patient Level Implementation Strategies:

Patients eligible for the patient level strategies must have had a recent visit at a participating clinic; are at least 18 years of age; currently use tobacco; live in a PP census tract; speak English or Spanish; have a valid cell phone number in the their clinics' EHR that can send and receive text messages; and have not opted out of the study. The patient level randomization is based on Quit Services response. Descriptions of the patient level conditions are as follows:

* Bundled: All patient level strategies will address the content of increasing reach of the Utah Tobacco Quit Services and SDOH.
* Non-Bundled: All patient level strategies will address only the content of increasing reach of the Utah Tobacco Quit Services.
* Reactive Patient Navigation Only (RPN): Patient can request to speak to a Community Health Worker (CHW), over 12 months following a patient's initial clinic visit, at any time.
* Proactive Patient Navigation (PPN): Patient is proactively called, over 12 months following a patient's initial clinic visit, by a CHW up to 4 times.
* Dose: The number of proactive outreach opportunities for Conversational Agent (CA) the patient receives. Patient will receive 1, 3, 6, 9, or 12 opportunities for CA, over 12 months following a patient's initial clinic visit, that includes a simple one-touch response to directly connect to the Quit Services or the CHW.

Eligible individuals who do not enroll in the Quit Services after four weeks will be randomly assigned to one of 20 conditions in the 2X2X5 factorial design (Non-Bundled & RPN & Dose, Non-Bundled & PPN & Dose, Bundled & RPN & Dose, Bundled & PPN & Dose, for each dose of 1, 3, 6, 9, 12).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Speak English or Spanish
* Currently use tobacco
* Live in a persistent poverty census tract
* Present at participating clinics
* Valid cell phone number in the electronic health record (EHR)
* Electronic health records indicate they have not opted out of receiving text contact from the clinic

Exclusion Criteria:

* Opt-out of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1560 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2027-11-15 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Reach of the Quit Services | up to 12 months after study enrollment
  Reach of the Quit Services is the number of eligible patients who officially enroll in the Quit Services over the total number of eligible patients.

SECONDARY OUTCOMES:
Association between patient and clinic level predictor variables | 12 Months
  We will perform separate analyses using generalized linear mixed models to investigate the association between patient and clinic level predictor variables (such as Reach, Effectiveness, Adoption, Implementation, and Maintenance.) derived from our conceptual model with process outcomes for AAC, CA, and PN dissemination and implementation strategies.
  This outcome measure will report if there is an associate between patient and clinical level predictor variable.
Reach -- SDOH | Up to 12 months after enrollment in study.
  Proportion of patients who use tobacco, are seen at a participating clinic, live in PP census tract, and receive services for SDOH (among sampled patients only)
Patient Abstinence | Up to 12 months after study enrollment
  Proportion of patients who report 7 or 30 day abstinence among those sampled.
Reach - Offer | Up to 12 months after study enrollment
  Proportion of patients offered connection to Quit Services/total patients offered connection to Quit Services.
Reach -- Connect | Up to 12 months after study enrollment
  Proportion of patients who accept connection to Quit Services out of eligible patients
Patient Engagement | Up to 12 months after study enrollment
  Proportion of patients who interact with CA or PN out of eligible patients.
Cost-Effectiveness | Up to 12 months after study enrollment
  Cost-effectiveness of strategies

CONTACTS AND LOCATIONS:
Overall Officials: Chelsey Schlechter, MPH, PhD, Principal Investigator — Huntsman Cancer Institute/ University of Utah
Locations (1):
- Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah, United States